CLINICAL TRIAL: NCT07243418
Title: Dual-cohort, Single-arm, Exploratory Phase II Clinical Study of Hetrombopag for Primary/Secondary Prevention of Thrombocytopenia Induced by ADC Drugs in Breast Cancer
Brief Title: Hetrombopag for the Prevention of ADC-Induced Thrombocytopenia in Breast Cancer: An Exploratory, Dual-Cohort, Phase 2 Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HQBP-BC-01
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: CTIT-Chemotherapy Induced Thrombocytopenia; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary prevention (Experimental)
  Interventions: Drug: herombopag olamine tablets
- Secondary prevention (Experimental)
  Interventions: Drug: herombopag olamine tablets

INTERVENTIONS:
Drug: herombopag olamine tablets — Starting from day 1 after chemotherapy, oral administration ofherombopag olamine tablets at a dose of 5mg per day (the initial dose) was administered for 14 consecutive days. Blood routine tests of the subjects were collected on days 7, 10, and 14 respectively, and the dose of herombopag olamine tablets was adjusted according to PLT

SUMMARY:
The title of this study is: A two-cohort, single-arm, exploratory Phase II clinical study on the primary/secondary prevention ADC drug of heltrombopag for thrombocytopenia caused by breast cancer. This study is a two-cohort, single-arm, open-label, exploratory clinical trial for the prevention of thrombocytopenia caused by ADC drug treatment for breast cancer. This research was supported by Fujian Cancer Hospital. The protocol has been reviewed by the Ethics Committee of Fujian Cancer Hospital, which has agreed to conduct this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 -75 years old, gender not limited.
* 2. Breast cancer patients diagnosed by histopathological or cytological examination;
* 3. Cohort 1: Planned to receive ADC drug treatment; Cohort 2: Patients who received ADC drug treatment in the previous chemotherapy cycle and had a minimum PLT value of less than 75*109/L are expected to maintain the same chemotherapy regimen for ≥2 cycles.
* 4. Expected survival period ≥12 weeks;
* 5. Physical condition ECOG PS score: 0-2 points;
* 6. The laboratory inspection indicators meet the following requirements:

  1. Renal function: Cr≤UNL (upper limit of normal) ×1.5, endogenous creatinine clearance rate (Ccr) ≥55 ml/min;
  2. Liver function: Total bilirubin ≤ULN×1.5; ALT and AST≤ULN×3; If it is intrahepatic cholangiocarcinoma or liver metastasis, the total bilirubin shall not exceed three times the upper limit of normal, and the transaminase shall not exceed five times the upper limit of normal.
  3. Coagulation function: The international normalized ratio of prothrombin time is ≤ULN×1.5, and some prothrombin times are within the normal range.
* 7. Women of childbearing age agree to use contraception during the study period and for six months after the end of the study. And not a lactating patient; Male patients who agreed to contraception during the study period and for 6 months after the end of the study;
* 8. Those who have not participated in other drug clinical trials within 4 weeks prior to enrollment;
* 9. The subjects can understand the situation of this study and voluntarily sign the informed consent form.
* 10. No serious complications such as active massive gastrointestinal bleeding, perforation, jaundice, gastrointestinal obstruction, or non-cancerous fever > 38℃;
* 11. Those with good expected compliance can follow up on the therapeutic effect and adverse reactions as required by the protocol.

Exclusion Criteria:

* 1. Screening or baseline platelet value ≤10×109/L;
* 2. Patients who are currently taking pyrotinib, dalciclib or other CDK4/6 class drugs
* 3. Thrombocytopenia caused by non-tumor treatment occurred within 6 months before screening, including but not limited to liver cirrhosis with hypersplenism, infection and bleeding, etc.
* 4. Suffering from other hematopoietic system diseases except for thrombocytopenia caused by anti-tumor therapy, including leukemia, primary immune thrombocytopenia, myeloproliferative disorders, multiple myeloma and myelodysplastic syndrome, etc.
* 5. Combined bone marrow invasion or bone marrow metastasis;
* 6. Had received radiotherapy for the pelvis, spine and bone irradiation within 3 months before screening:
* 7. Any history of arterial or venous thrombosis within 6 months prior to the screening;
* 8. There were severe clinical manifestations of bleeding (such as gastrointestinal bleeding, etc.) within 2 weeks before screening;
* 9. Patients with severe cardiovascular diseases (such as NYHA cardiac function score III-IV), arrhythmias known to increase the risk of thromboembolism such as atrial fibrillation, after coronary stent implantation, angioplasty, and after coronary artery bypass grafting within 6 months prior to screening;
* 10. Brain tumors or brain metastases;
* 11. When the absolute value of neutrophils is less than 1.0×109/L and hemoglobin is less than 80g/L, the use of granulocyte colony-stimulating factor and red blood cell, EPO infusion therapy that conforms to clinical routine is allowed.
* 12. Significantly abnormal liver function: For patients without liver metastasis, ALT/AST > 3ULN (upper limit of normal value), and TBIL > 3ULN; Patients with liver metastasis have ALT/AST≥5ULN and TBIL≥5ULN.
* 13. Abnormal renal function: Serum creatinine ≥1.5ULN or eGFR≤60 ml/min (Cockcroft-Gault formula)
* 14. Platelet transfusion was received within 2 days before enrollment;
* 15. Received treatment with human recombinant thrombopoietin (rhTPO), human recombinant interleukin-11 (rhIL-11), or thrombopoietin receptor agonists (such as eltrombopag, avatracopag) within 10 days before screening;
* 16. Patients who are known or expected to be allergic to or intolerant to the active ingredients or excipients of heltrombopag ethanolamine tablets (excipients include: cellulose-lactose, low-substitution hydroxypropyl cellulose, magnesium stearate, film-coated premixes);
* 17. Pregnant or lactating women;
* 18. Those who were considered unsuitable for inclusion by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of Grade 3 and above Cancer Therapy - Induced Thrombocytopenia (CTIT) | During the period of oral medication (14 days

IPD SHARING:
Plan to Share IPD: No